CLINICAL TRIAL: NCT01787604
Title: Superiority Trial of Aortic Root Reimplantation Procedure Versus Aortic Valve Reimplantation Procedure
Brief Title: Study of Aortic Root Reimplantation Procedure
Acronym: STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Principal Investigator, Dmitry Khvan, cardiac surgeon, Meshalkin Research Institute of Pathology of Circulation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STAR
Record Dates: First submitted 2013-01-30; First posted 2013-02-08 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-03

CONDITIONS: Ascending Aortic Aneurism; Aortic Valve Insufficiency
Keywords: Valve-sparing; Valve repair
MeSH Terms: conditions — Aortic Valve Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aortic Root Reimplantation Procedure (Active Comparator): Aortic Root Reimplantation Procedure
  Interventions: Procedure: Aortic Root Reimplantation Procedure
- Aortic Valve Reimplantation Procedure (Active Comparator): Aortic Valve Reimplantation Procedure
  Interventions: Procedure: Aortic Valve Reimplantation Procedure

INTERVENTIONS:
Procedure: Aortic Root Reimplantation Procedure — Modified Florida Sleeve.
  Other Names: Modified Florida Sleeve.
  Arms: Aortic Root Reimplantation Procedure
Procedure: Aortic Valve Reimplantation Procedure — David I
  Other Names: David I
  Arms: Aortic Valve Reimplantation Procedure

SUMMARY:
Authors hypothesize that aortic root reimplantation procedure is superior over standard aortic valve reimplantation procedure in the incidence of aortic valve replacement.

DETAILED DESCRIPTION:
A single blind prospective randomized superiority study is conducted. Our hypothesis is that there is difference in the incidence of aortic valve replacement between the standard aortic valve reimplantation procedure and aortic root reimplantation procedure more than 21.1%. If there is truly difference between groups (Aortic Root Reimplantation Procedure and Aortic Valve Reimplantation Procedure), then total 64 patients for both groups are required to be 80% sure that the upper limit of a one-sided 95% confidence interval would reveal a difference in favour of the Aortic Root Reimplantation Procedure of 21.1%. The blinding process is applied to a patient, who is informed about received valve-sparing operation, but don't know the type of the last. The study was approved by Institutional Review Board. Depending on a type of the procedure, the patients are divided into two groups: Aortic Root Reimplantation Procedure group includes 32 patients and Aortic Valve Reimplantation Procedure group consists of 32 patients. Randomization is conducted intraoperatively by using accidental sampling after examining the aortic valve and making a decision on the possibility of a valve-sparing operation.

ELIGIBILITY:
Inclusion Criteria:

* Aortic insufficiency 2+
* Ascending aorta or aortic root of greater than 4.5 cm (> 4.0 cm in Marfan syndrome)
* Good conditions of aortic cusps

Exclusion Criteria:

* Aortic annulus more than 32 mm
* Aortic cusps destruction
* Critical aortic cusps elongation
* Aortic root dissection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2015-11-20 (Actual); Study Completion 2015-11-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Meshalkin State Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- [Result] Alexander Chernyavskiy, Sergey Alsov, Dmitry Khvan, Dmitry Sirota. Extravalvular exoprosthetic repair of aortic root: first experience. Kardiochirurgia i Torakochirurgia Polska 2012; 9 (4): 409-414 DOI: 10.5114/kitp.2012.32675
- [Result] Чернявский А. М., Хван Д. С., Альсов С. А., Сирота Д. А., Ляшенко М. М. Результаты реимплантации корня аорты в протез у пациентов с аневризмой восходящего отдела аорты и недостаточностью аортального клапана. Патология кровообращения и кардиохирургия. 2015;19(4):38-47. http://dx.doi.org/10.21688/1681-3472-2015-4-38-47

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aortic Root Reimplantation Procedure | Aortic Valve Reimplantation Procedure
Started | 32 | 32
Completed | 28 | 28
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aortic Root Reimplantation Procedure | Aortic Valve Reimplantation Procedure | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [52 to 65] | 56 [50 to 63] | 58 [52 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 25 | 25 | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Aortic Insufficiency More Than 2+ (Percentage, Kaplan-Meier)
Description: Estimated percentage of participants free from aortic insufficiency (AI) more than 2+ measured by echocardiography for a 4 years after treatment..
Time Frame: up to 4 yeras
Measure: Number; unit: percentage of participants
Arm/Group | Aortic Root Reimplantation Procedure | Aortic Valve Reimplantation Procedure
Number analyzed (Participants) | 32 | 32
percentage of participants | 88.2 | 87.7

2. Secondary Outcome: Survival (Percentage, Kaplan-Meier)
Description: Estimated percentage of alive participants for 4 years after treatment.
Time Frame: up to 4 yeras
Measure: Number; unit: percentage of participants
Arm/Group | Aortic Root Reimplantation Procedure | Aortic Valve Reimplantation Procedure
Number analyzed (Participants) | 32 | 32
percentage of participants | 82.7 | 84.6

ADVERSE EVENTS:
Time Frame: up to 4 yeras
Arm/Group | Aortic Root Reimplantation Procedure | Aortic Valve Reimplantation Procedure
All-Cause Mortality (participants affected / at risk) | 4/32 | 4/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes